CLINICAL TRIAL: NCT06320574
Title: Nurses' Competence for Bedside Ultrasound Assessment of Gastric Content: a Cohort Study
Brief Title: Nurses' Competence in Gastric Ultrasound
Acronym: SKILLS-1
Status: Not yet recruiting | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-16880
Record Dates: First submitted 2024-02-11; First posted 2024-03-20 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-02

CONDITIONS: Gastric Content; Healthy Volunteers
Keywords: Gastric Ultrasound; Nurses; Training; Competency; point-of-care ultrasound

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational cohort study is to investigate gastric ultrasound skills in surgical nurses. The main question it aims to answer is:

• how much training is required for surgical nurses to obtain competency in performing gastric ultrasound.

Participants will follow a training involving

* theoretical background using e-learning, picture library and lecture
* practical skill development in an interactive hands-on workshop on live models directed by expert gastric ultrasonographer
* and formative assessments during training sessions scanning healthy volunteers by participants and examiners (expert gastric ultrasonographers).

DETAILED DESCRIPTION:
Aims: To determine the amount of training bachelor nurses require to achieve competence in the bedside point-of-care ultrasound technique for qualitative assessment of gastric content.

Study design: prospective cohort educational study

Study population: The participants are six nurses at bachelor level with at least 1 year of experience with surgical patients. Volunteers are healthy persons without a pre-existing abnormal anatomy of the upper gastrointestinal tract.

Main study parameters/endpoints Primary outcome is the number of ultrasound examinations which is required to achieve competence in the performance of ultrasonography qualitative assessment of gastric content. The number of ultrasound assessments nurses need to achieve 90% success rate in 10 consecutive ultrasound assessments among healthy volunteers. Reference test is the ultrasound assessment of examiners experienced in (gastric) ultrasound.

Methods: The education program is developed according to relevant literature, panel discussion of a project group including relevant experts on gastric ultrasonography and nursing education.

Six nurses will follow the education program including didactic teachting and formal assessments. The didactic teaching include1) theoretical background using e-learning, picture library and lecture and 2) practical skill development in an interactive hands-on workshop on live models directed by expert gastric ultrasonographer. Formative assessments will be done by scanning healthy volunteers by participants and examiners (expert gastric ultrasonographers). Volunteers will be asked to adhere to a randomized prandial. Participants and examiners will be blinded for the prandial status of the volunteer.

Analysis: Cumulative sum scores will be estimated to determine the number of trainings that is required.

ELIGIBILITY:
Inclusion criteria for nurses:

* nurses with at least 1 year experience at the unit;
* nurses with a bachelor's degree in nursing;
* nurses with a particular interest in ultrasonography.
* nurses without previous experience in ultrasonography;

Inclusion criteria for healthy volunteers:

* no history of abnormal anatomy or surgery of the upper gastro-intestinal tract (previous oesophageal-, gastric-, or upper abdomen surgery, or hiatus hernia);
* no diabetes mellitus

Exclusion criteria

• subjects who do not provide written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Nurses employed at the gastro-intestinal and oncology department in the Radboudumc who underwent G-POCUS training The training goals are sufficient knowledge, skills, and attitude to achieve sufficient competence. The course will be divided into three components: 1) didactic teaching in an e-learning, study material, and picture library; 2) Interactive session consisting of a hands-on workshop by the expert sonographer and scanning of other trainees; 3) performing G-POCUS in healthy volunteers in a training environment with formal assessment.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Estimated)
Dates: Start 2024-03-14 (Estimated); Primary Completion 2024-04-20 (Estimated); Study Completion 2024-08-01 (Estimated)

PRIMARY OUTCOMES:
Number of required training | 5 days of ultrasound assessment of 6 volunteers will be performed in 2 kind of prandial status (leading to 12 assessment per day)
  Main study endpoint was the number of scans nurses require to achieve sufficient competency in gastric ultrasound assessment. Competence was defined as 90% success rate in the 10 consecutive gastric ultrasound assessments.

CONTACTS AND LOCATIONS:
Overall Officials: Getty Huisman-de Waal, PhD, Principal Investigator — Radboud University Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bouvet L, Mazoit JX, Chassard D, Allaouchiche B, Boselli E, Benhamou D. Clinical assessment of the ultrasonographic measurement of antral area for estimating preoperative gastric content and volume. Anesthesiology. 2011 May;114(5):1086-92. doi: 10.1097/ALN.0b013e31820dee48. PMID 21364462
- [Background] Perlas A, Arzola C, Van de Putte P. Point-of-care gastric ultrasound and aspiration risk assessment: a narrative review. Can J Anaesth. 2018 Apr;65(4):437-448. doi: 10.1007/s12630-017-1031-9. Epub 2017 Dec 11. PMID 29230709
- [Background] Perlas A, Van de Putte P, Van Houwe P, Chan VW. I-AIM framework for point-of-care gastric ultrasound. Br J Anaesth. 2016 Jan;116(1):7-11. doi: 10.1093/bja/aev113. Epub 2015 May 7. No abstract available. PMID 25951832
- [Background] Lamm R, Collins M, Bloom J, Joel M, Iosif L, Park D, Reny J, Schultz S, Phillips B, Schwenk E, Costanzo C. Novice User Learning Curve for Handheld Gastric Point of Care Ultrasound Evaluations to Detect Delayed Return of Postoperative Peristalsis. Am Surg. 2023 Dec;89(12):6290-6292. doi: 10.1177/00031348231156770. Epub 2023 Feb 14. No abstract available. PMID 36787243
- [Background] Arzola C, Carvalho JC, Cubillos J, Ye XY, Perlas A. Anesthesiologists' learning curves for bedside qualitative ultrasound assessment of gastric content: a cohort study. Can J Anaesth. 2013 Aug;60(8):771-9. doi: 10.1007/s12630-013-9974-y. Epub 2013 May 24. PMID 23703533
- [Background] Brotfain E, Erblat A, Luft P, Elir A, Gruenbaum BF, Livshiz-Riven I, Koyfman A, Fridrich D, Koyfman L, Friger M, Grivnev A, Zlotnik A, Klein M. Nurse-performed ultrasound assessment of gastric residual volume and enteral nasogastric tube placement in the general intensive care unit. Intensive Crit Care Nurs. 2022 Apr;69:103183. doi: 10.1016/j.iccn.2021.103183. Epub 2021 Dec 16. PMID 34924254